CLINICAL TRIAL: NCT02000375
Title: A Phase II Non Randomized Study Evaluating the Role of Androgen Receptors as Targets for Therapy of Pre-treated Post-menopausal Patients With ER/PgR-negative/AR-positive or ER and/or PgRpositive/ AR-positive Metastatic Breast Cancer (ARTT)
Brief Title: A Phase II Study Evaluating the Role of Androgen Receptors as Targets for Therapy of Pre-treated Post-menopausal Patients With ER/PgR-negative/AR-positive or ER and/or PgRpositive/ AR-positive Metastatic Breast Cancer (ARTT)
Acronym: ARTT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow recruitment and recent new published data
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST174.08; 2012-003510-13 (EudraCT Number)
Record Dates: First submitted 2013-11-21; First posted 2013-12-04 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Metastatic Breastcancer; Estrogen Receptor Positive Breast Cancer; Estrogen Receptor Negative Neoplasm; Progesterone Receptor Positive Tumor; Progesterone Receptor Negative Neoplasm; Androgen Receptor Gene Overexpression
Keywords: metastatic breastcancer; ER/PgR-negative/AR-positive; ER and/or PgR-positive/AR-positive; Androgen Receptor positve
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DHEA (Experimental): Daily oral administration of DHEA at the dosage of 100 mg/die in combination with a daily oral administration of anastrozole at dosage of 1 mg/die or letrozole at the dosage of 2.5 mg/die or exemestane at the dosage of 25 mg/die without interruption.
  Interventions: Drug: DHEA

INTERVENTIONS:
Drug: DHEA — DHEA: Daily oral administration of DHEA(Dehydroepiandrosterone) at the dosage of 100 mg/die in combination with a daily oral administration of anastrozole at dosage of 1 mg/die or letrozole at the dosage of 2.5 mg/die or exemestane at the dosage of 25 mg/die without interruption.
  Other Names: Dehydroepiandrosterone

SUMMARY:
A phase II non randomized study evaluating the role of Androgen Receptors as Targets for therapy of pre-treated postmenopausal patients with ER/PgR-negative/AR-positive or ER and/or PgR-positive/AR-positive metastatic breast cancer.

Study Design: Multicentric, Open-label not randomized trial.

Description of Study Treatment:

Daily oral administration of DHEA (Dehydroepiandrosterone) at the dosage of 100 mg/die in combination with a daily oral administration of anastrozole at dosage of 1 mg/die or letrozole at the dosage of 2.5 mg/die or exemestane at the dosage of 25 mg/die without interruption until discontinuation for progression of disease, unacceptable toxicity or discontinuation/withdrawal of participants from study treatment.

Number of Subjects:

12 patients per group in the first step; if the number of responders is greater or equal to 2, recruitment will continue up to a total of 35 patients (per group).

For the biological part, we will evaluate:

1. Correlation between AR expression and clinical and biological features (tumor size, nodal status, histotype, grading, proliferative index, ER, PgR, HER2)
2. Evaluation of AR expression on primitive and/or metastatic site in the two distinct populations of patients: ER/PgR- negative/ARpositive and ER-positive and/or PgR-positive/AR-positive
3. Evaluation of ER, PgR, HER2 expression on tumor cells of metastatic site (when it is possible) and comparison with the same features of primitive tumor.
4. CTCs analysis in term of molecular characteristics (gene expression and mutations) and functionality (vitality and tumorigenicity).
5. Prognostic and predictive role of Circulating Tumor Cells (CTC) evaluated at baseline before study treatment and at the moment of discontinuation of treatment.

DETAILED DESCRIPTION:
A phase II non randomized study evaluating the role of Androgen Receptors as Targets for therapy of pre-treated postmenopausal patients with ER/PgR-negative/AR-positive or ER and/or PgR-positive/AR-positive metastatic breast cancer.

Study Design: Multicentric, Open-label not randomized trial.

Description of Study Treatment:

Daily oral administration of DHEA (Dehydroepiandrosterone) at the dosage of 100 mg/die in combination with a daily oral administration of anastrozole at dosage of 1 mg/die or letrozole at the dosage of 2.5 mg/die or exemestane at the dosage of 25 mg/die without interruption until discontinuation for progression of disease, unacceptable toxicity or discontinuation/withdrawal of participants from study treatment.

Number of Subjects:

12 patients per group in the first step; if the number of responders is greater or equal to 2, recruitment will continue up to a total of 35 patients (per group).

For the biological part, we will evaluate:

1. Correlation between AR expression and clinical and biological features (tumor size, nodal status, histotype, grading, proliferative index, ER, PgR, HER2)
2. Evaluation of AR expression on primitive and/or metastatic site in the two distinct populations of patients: ER/PgR- negative/ARpositive and ER-positive and/or PgR-positive/AR-positive
3. Evaluation of ER, PgR, HER2 expression on tumor cells of metastatic site (when it is possible) and comparison with the same features of primitive tumor.
4. CTCs analysis in term of molecular characteristics (gene expression and mutations) and functionality (vitality and tumorigenicity).
5. Prognostic and predictive role of Circulating Tumor Cells (CTC) evaluated at baseline before study treatment and at the moment of discontinuation of treatment.

Statistical Considerations:

The sample size required for each treatment arm will be predicted using a SIMON two-stage design with a 10 percent alpha and beta error.

Assuming an acceptable minimum clinical benefit P0 equal to 10 percent and an auspicious clinical benefit P1 equal to 30 percent, we plan to recruit 12 patients per group in the first step.

If the number of responders is greater or equal to 2, recruitment will continue up to a total of 35 patients (per group).

If the number of responders is greater or equal to 6, the combination will be considered active and worthy of further evaluation.

If a subgroup population is discontinued at the end of the first step, the study will be continued with the other subgroup.

ELIGIBILITY:
Inclusion Criteria:

1. Histological-documented diagnosis of invasive breast cancer.
2. Clinical diagnosis of metastatic breast cancer.
3. AR receptor positivity of primary tumor cells or tumor cells of a metastatic site is required. It is strongly recommended that 4 unstained and freshly cut 3-4 μ slides from the primary tumor (or metastatic if the primary is not available) be submitted for IRCCS IRST Laboratorio di Bioscienze for confirmation of AR eligibility; however, if that is not possible, a formalin-fixed paraffin-embedded (FFPE) tissue block will be submitted .

   Tumors with ≥10% positively nuclear-stained cells by immunohistochemistry (IHC) are considered positive for AR.
4. Primary tumor cells or tumor cells of a metastatic site can be ER-positive and/or PgRpositive or ER-negative/PgR-negative . Hormone receptor positivity is defined as ER and/or PgR greater than 10 fmol/mg by biochemical assay or greater or equal than 10 percent positive cells by immunohistochemistry.
5. Primary tumor cells or tumor cells of a metastatic site must be HER2 negative.
6. Measurable disease, defined in accord to RECIST criteria (version 1.1) as

   1. at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with CT scan or MRI (if slice thickness no grater than 5 mm. If slice thicknesses grater than 5 mm the minimum size miserable lesions at baseline should be twice the slice thickness of baseline scans)
   2. to be considered pathologically enlarged and measurable, a lymph node must be ≥ 15 mm in short axis when assessed by CT scan or MRI (if slice thickness no grater than 5 mm. If slice thicknesses grater than 5 mm the minimum size miserable nodes at baseline).
7. In case of ER-pos disease, previous endocrine treatment in adjuvant or metastatic setting is required and patients must be resistant to aromatase inhibitors that means:

   * AI in adjuvant setting: patients should have been treated for at least 1 year and have had a recurrence during this treatment or in the first year after finishing adjuvant treatment
   * AI in advanced disease: patients must have received the AI lasting at least 6 months, during which patients must have achieved a tumor response or stabilization ,and have had an objective progression during treatment
8. No more than 2 previous lines of chemotherapy for ER-pos tumors and not more than 3 lines of chemotherapy for ER-neg tumors are allowed
9. Post-menopausal status defined as:

   1. Patients of any age who have had a bilateral oophorectomy (including radiation castration)
   2. Patients 56 years old or older. If the patient has any evidence of ovarian function, biochemical evidence of definite postmenopausal status (defined as estradiol, LH, and FSH in the postmenopausal range) is required.
   3. Patients 55 years old or younger without period in the last 12 month or with biochemical evidence of definite postmenopausal status (defined as estradiol, LH, and FSH in the postmenopausal range).
10. At least 18 years of age
11. Life expectancy greater of 12 weeks
12. ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2
13. Adequate organ and marrow function as defined below:

    * leukocytes >3,000/mL
    * absolute neutrophil count >1,500/mL
    * platelets >100,000/mL
    * total bilirubin within normal institutional limits
    * AST(SGOT)/ALT(SGPT) <2.5 X institutional ULN
    * creatinine within normal institutional limits OR
    * creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
14. Patients must exhibit capability of swallow tablets
15. Patients must exhibit compliance with an oral treatment
16. Patients must exhibit geographic proximity that allows regular access to the Institute for clinical and instrumental examinations is required
17. Participants must be willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. AR-receptor negativity of primary tumor cells or tumor cells of a metastatic site. AR is reported as negative if less than 10% of cells immunostained in a tumor.
2. HER2 positivity of primary tumor cells or tumor cells of a metastatic site
3. Physician opinion of a too rapid disease progression (like disease widespread in visceral organs like liver or lung in few months) that could suggest the physician a more benefit from chemotherapy treatment even if eligibility criteria for enrollment are satisfied
4. Chemotherapy administration within 3 weeks prior to start of protocol therapy or not recovered from adverse events due to agents administered more than 3 weeks earlier
5. Brain metastasis not treated or in progression requiring treatment (radiotherapy, surgery or high dose steroidal and antiedemigen treatment) in the 2 weeks prior to start of protocol therapy. Patients with brain metastasis as unique site of metastasis are excluded
6. Have received supplement of estrogen or progesterone within 4 weeks prior to study enter
7. Major surgery during the 21 days before before starting of protocol therapy or planned during the study treatment
8. Other detectable malignant neoplastic diseases (even a second primitive breast cancer) in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma of the skin and in situ carcinoma of the uterine cervix)
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
10. Participation in another clinical trial with any investigational agents within 3 weeks prior to study screening
11. Previous treatment with androgens or DHEA. Previous treatment with AI is required in case of ER+ and/or PgR positive tumors
12. History of allergic reactions attributed to compounds of similar chemical or biologic composition to DHEA or AI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate (CB) | 36 months
  the proportion of patients with stability, partial response and complete response of the disease after 4 months of therapy.

SECONDARY OUTCOMES:
Time to tumor progression (TTP) | 36 months
  It is defined as the time from randomization until objective tumor progression NOT including death.
Duration of response (DOR) | 36 months
  The time from the date of response documentation to the date of disease progression documentation.
Overall survival (OS) | 36 months
  The time from the date of randomization to date of death from any cause.
Quality of life Quality of life Quality of life Quality of life | 36 months
  FACT ( Functional Assessment of Cancer Therapy ) -B : a 36-item compilation, subdivided into four primary QOL (Quality of life) domains and a disease specific domain - additional concerns for breast cancer.
Correlation between AR expression and clinical and biological features | 36 months
  Immunohistochemistry for steroid receptors. Antigen expression is evaluated at light microscope (x 200) by two independent observers.
  The positivity is expressed as the percentage ratio between immunoreactive and total number of tumor cells. The cut off value > 10%for AR will be adopted.
Evaluation of AR expression on primitive and/or metastatic site in the two distinct populations of patients ( ER/PgR- negative/ARpositive and ER-positive and/or PgR-positive/AR-positive) | 36 months
  Immunohistochemistry for steroid receptors. Antigen expression is evaluated at light microscope (x 200) by two independent observers.
  The positivity is expressed as the percentage ratio between immunoreactive and total number of tumor cells. The cut off value > 10%for AR will be adopted.
Evaluation of ER, PgR, HER2 expression on tumor cells of metastatic sites (when it is possible) and comparison with the same features of the the primary site. | 36 months
  Immunohistochemistry for steroid receptors. Antigen expression is evaluated at light microscope (x 200) by two independent observers.
  The positivity is expressed as the percentage ratio between immunoreactive and total number of tumor cells. The cut off value > 10%for AR will be adopted.
Circulating Tumor Cells (CTCs) analysis [Optionally, only for patients enrolled at IRCCS IRST of Meldola and who signed additional informed consent ] | 36 months
  Analyzing 15-20 ml peripheral blood (PB). The blood collection will be taken before starting treatment at baseline and at the end of treatment.
Safety | 36 months
  Assessed by collecting adverse events (AE) and serious adverse events (SAE) during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Pietri, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (8):
- Italy (8):
  - Irccs Irst, Meldola, FC
  - Oncologia medica , PO FAENZA, Ausl della Romagna, Faenza, RA
  - Oncologia Medica PO Lugo, AUSL della Romagna, Lugo, RA
  - Oncologia medica PO Ravenna AUSL della Romagna, Ravenna, RA
  - Oncologia Medica PO Cattolica AUSL della Romagna, Cattolica
  - Oncologia Medica,E.O. Ospedali Galliera, Genova
  - Oncologia Medica AOU Policlinico di Modena, Modena
  - Oncologia medica PO Rimini AUSL della Romagna, Rimini

REFERENCES:
- [Derived] Pietri E, Massa I, Bravaccini S, Ravaioli S, Tumedei MM, Petracci E, Donati C, Schirone A, Piacentini F, Gianni L, Nicolini M, Campadelli E, Gennari A, Saba A, Campi B, Valmorri L, Andreis D, Fabbri F, Amadori D, Rocca A. Phase II Study of Dehydroepiandrosterone in Androgen Receptor-Positive Metastatic Breast Cancer. Oncologist. 2019 Jun;24(6):743-e205. doi: 10.1634/theoncologist.2018-0243. Epub 2018 Dec 27. PMID 30591548